CLINICAL TRIAL: NCT04317898
Title: Ultrasound-Guided Serratus Plane Block Vs Paravertebral Block For Chronic Post-mastectomy Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Abo eldahab Ali elden, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: analgesia in chronic PMPs
Record Dates: First submitted 2020-03-20; First posted 2020-03-23 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Post-mastectomy Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- serratus plane block (Active Comparator): 20 ml of Bupivacine 0.25% +80mg triamcinlone will be injected in serratus plane under ultrasound.
  Interventions: Procedure: serratus plane block by ultra-sound
- paravertebral block (Active Comparator): 10 ml of bubivacine 0.25% +80 mg triamcinlone will be injected at T2 level (paravertebral) under ultrasound.
  Interventions: Procedure: paravertebral block by ultra-sound

INTERVENTIONS:
Procedure: serratus plane block by ultra-sound — To perform Serratus block, patients will be placed in the lateral decubitus position with the affected side facing up, or in the prone position with the affected side facing the operator . After sterile preparation, a linear ultrasound probe will be utilized to identify the latissimusdorsi and serratus anterior muscles in a sagittal plane. The plane superficial to the serratus anterior muscle and below the latissimusdorsi muscle will be identified. The skin will be topicalized with 1 mL of 1% lidocaine using a 30-gauge needle. Using an in-plane approach, a 25-gauge 1.5-cm needle will be used to inject a total of 20-mL of 0.25% bupivacaine with 80 mg of triamcinlone under direct ultrasound visualization.
  Arms: serratus plane block
Procedure: paravertebral block by ultra-sound — TPVB will be given using high frequency linear US transducer, place the probe parallel to the vertebral spine at T2 level and shifted 2-3 cm laterally to obtain the appropriate visualization. Following the identification of plura, transverse process and paravertebral space, the needle will be inserted in caudocranial direction using in-plane approach. Confirm negative vessel or pleural breach via aspiration then proceed with local anaesthetic 10ml of 0.25% bubivacine and 80mg triamcinlone slowly; the pleura will be seen to be pushed downward.
  Arms: paravertebral block

SUMMARY:
compare the analgesic efficacy between ultrasound paraverbral block and serratus block in post mastectomy pain.

DETAILED DESCRIPTION:
It is reported that postmastectomy pain syndrome (PMPS) is a common problem, ranging from 25% to 60%.

The pain is localized in the axilla, medial upper arm, breast, and/or chest wall and lasting beyond three months after surgery when all other causes of pain such as infection have been eliminated.

The pain seriously affects the patient's mood, everyday activities, and social function and causes heavy economic burden for the healthcare system.

Postmastectomy pain syndrome (PMPS) itself is not a specific diagnosis but rather describes a cluster of symptoms frequently observed in breast cancer survivors following treatment.

Many patients will experience short-term nociceptive pain after breast cancer treatment. However, with PMPS, patients frequently experience persistent neuropathic-type pain: burning, tingling, aching, a subjective sense of "tightness" around the chest wall, or even phantom breast or nipple pain. Neuropathic pain results from dysfunction of the peripheral nerves caused by surgery, radiation, or neurotoxic chemotherapies.

Currently, there are a wide variety of approaches to treat this type of pain. physical therapy has been employed as a modality to improve physical function.

As far as interventional procedures, intercostal nerve blockade, stellate ganglion blockade, and paravertebral blockade have all been utilized with varying degrees of success.

Paraverberal blocks have superseded thoracic epidurals when it comes to choice of a regional anaesthesia technique to provide analgesia for breast surgery.

The injection of local anaesthetic solution in the paravertebral space results in a unilateral block, which is sensory, motor, and sympathetic. The uptake of the local anaesthetic solution is enhanced due to the absence of fascial sheaths binding the spinal nerves.

Another potential target for an interventional procedure for chronic pain after treatment for breast cancer is the serratus plane. The serratus plane block is a novel ultrasound-guided nerve block, which is able to anesthetize the hemithorax.

The serratus plane block relies on the fact that there are branches of the intercostal nerves following within 2 potential spaces, one superficial and one deep, surrounding the serratus anterior muscle. The serratus anterior muscle arises as strips from the first 9 ribs and converges posteriorly on the scapula to form the medial wall of the axilla.

The innervation of the serratus anterior muscle is via the long thoracic nerve (Bell's nerve), and the nerve itself is covered by the fascia of the serratus anterior muscle and lies anterior to the muscle.

ELIGIBILITY:
Inclusion Criteria:

* Patients have postmastectomy pain of neuropathic nature, DN4

  * 4 for at least 3ms duration.
* The intensity of postmastectomy pain on VAS score ≥ 5.
* Unsatisfactory treatment with 1st line antineuropathic drugs, Pregabalin(150 mg daily) or Deloxetine(60mg daily).

Exclusion Criteria:

* Infection of the skin at or near site of needle puncture.
* Coagulopathy .
* Drug hypersensitivity or allergy to the studied drugs.
* Central or peripheral neuropthy .
* Significant organ dysfunction .
* Morbid obesity (BMI>35kg/m2) .
* Vertebral anomalies.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients gaining ≥ 50% pain reduction at VAS Score from baseline value. | baseline
  Compare the analgesic efficacy between ultrasound paraverbral block and serratus block in chronic postmastectomy pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Mohammed Abd El-Latif, Prof of Anesthesia, Study Director — Mohammed MohammedAbd El-Latif; Ashraf Amin Mohammed, Prof of Anesthesia, Study Director — Ashraf Amin Mohammed; Rania Mohammed Abd El-Emam, Lecturer of Anesthesia, Study Director — Rania Mohammed Abd El-Emam

REFERENCES:
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Smith WC, Bourne D, Squair J, Phillips DO, Chambers WA. A retrospective cohort study of post mastectomy pain syndrome. Pain. 1999 Oct;83(1):91-5. doi: 10.1016/s0304-3959(99)00076-7. PMID 10506676
- [Background] Couceiro TC, Menezes TC, Valenca MM. Post-mastectomy pain syndrome: the magnitude of the problem. Rev Bras Anestesiol. 2009 May-Jun;59(3):358-65. doi: 10.1590/s0034-70942009000300012. English, Portuguese. PMID 19488550
- [Background] Peuckmann V, Ekholm O, Rasmussen NK, Groenvold M, Christiansen P, Moller S, Eriksen J, Sjogren P. Chronic pain and other sequelae in long-term breast cancer survivors: nationwide survey in Denmark. Eur J Pain. 2009 May;13(5):478-85. doi: 10.1016/j.ejpain.2008.05.015. Epub 2008 Jul 16. PMID 18635381
- [Background] Fernandez-Lao C, Cantarero-Villanueva I, Fernandez-de-Las-Penas C, del Moral-Avila R, Castro-Sanchez AM, Arroyo-Morales M. Effectiveness of a multidimensional physical therapy program on pain, pressure hypersensitivity, and trigger points in breast cancer survivors: a randomized controlled clinical trial. Clin J Pain. 2012 Feb;28(2):113-21. doi: 10.1097/AJP.0b013e318225dc02. PMID 21705873
- [Background] Wijayasinghe N, Andersen KG, Kehlet H. Neural blockade for persistent pain after breast cancer surgery. Reg Anesth Pain Med. 2014 Jul-Aug;39(4):272-8. doi: 10.1097/AAP.0000000000000101. PMID 24918332